CLINICAL TRIAL: NCT01339130
Title: Assessment of Social-emotional Functioning in Stroke, Frontotemporal Dementia, Alzheimer and Parkinson Diseases
Brief Title: Assessment of Social-emotional Functioning in Neurological Diseases
Acronym: Emotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI09-PR-GODEFROY; 2009-A00596-51 (Other: CHU)
Record Dates: First submitted 2011-03-31; First posted 2011-04-20 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Alzheimer Disease; Stroke; Parkinson's Disease; Lewy Body Dementia; Huntington Disease
Keywords: Alzheimer disease; Stroke; Frontotemporal Lobar Degeneration; Lewy Body Dementia; Huntington Disease; mild cognitive impairment; vascular injury; Parkinson's disease
MeSH Terms: conditions — Alzheimer Disease; Stroke; Parkinson Disease; Lewy Body Disease; Huntington Disease; Frontotemporal Lobar Degeneration; Cognitive Dysfunction; Vascular System Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- behavioral and physiological tests (Other): Computerized tests and Electrophysiological measurements
  Interventions: Behavioral: Computerized tests and Electrophysiological measurements

INTERVENTIONS:
Behavioral: Computerized tests and Electrophysiological measurements — * Computerized tests: used to evaluate the empathy The participant observes a computer screen on which appears different types of images or words that can evoke an emotion. The participant responds by pressing the screen with his finger. This is a choice between several answers and respond as quickly as possible.
  * Electrophysiological measurements: provide a measure of autonomic response to emotional stimuli: galvanic response (GSR) and electromyographic activity (EMG) of facial muscles (corrugator supercilii and zygomatic major).
  * Neuropsychological assessment includes an assessment of intellectual efficiency, perceptual and visual-constructive abilities, memory, executive and an assessment of behavior and mood from questionnaires.

SUMMARY:
Empathy, defined as the ability to understand others emotions, is a fundamental concept in social interactions. It is a psychological phenomenon involving various separable components : (i) the ability to feel and imagine the emotions, (ii) the ability to adopt the perspective of other people. Several neurological diseases with behavioral disorders may lead to impaired processing of social and/or emotional informations. These pathologies are likely to induce a lack of empathy that may result from impairments at different levels.

The objective is simply to study how others' emotions are understood and how this allows for regulation of personal behavior. This study is being carried out among patients seen for various health problems and who can make behavior changes. This study could help to understand some neurological diseases and thereby to identify them earlier and/or to better differentiate them.

DETAILED DESCRIPTION:
Empathy is a fundamental concept in social interactions, whose function is to understand the emotions felt by others. According to De Waal (2008), it is a multidimensional concept that involves two processes :(i) a system of emotional contagion or affective resonance (the unconscious and automatic sharing of the emotion of others) that establishes the emotional component of empathy, (ii) the ability to take perspective, that is the ability to imagine the subjective world of the other distinguishing oneself from him, forming the cognitive component of empathy.

Several neurological diseases with behavioral disorders may lead to impaired processing of social and/or emotional information. These pathologies are likely to induce a lack of empathy that may result from impairments at different levels.

The main objective of this study is to examine empathy in patients suffering from stroke (various locations with an emphasis on frontal stroke), Fronto-temporal dementia, Alzheimer and Parkinson diseases. The final assessment criterion is the overall score on the scale of empathy.

The patient will firstly receive a medical examination and clinical data are collected (past medical history, clinical neurological examination, diagnosis, description of first symptoms, course, current treatments)and brain imaging data. After checking inclusion criteria, information letter and the consent form will be returned.

The second visit will consist in neuropsychological assessment: general intellectual efficiency, perceptual and visual-constructive abilities, memory, executive and an assessment of behavior and mood from questionnaires The third and final visit will allow passing experimental tests. The experimental part will include the following tests: (1) recognition of emotional facial expressions; (2) tasks of theory of mind ; (3) task of empathy for pain.

A control group will also perform the neuropsychological and experimental tests.

The duration of the study participation for eligible patients and controls will vary according to the delay between each visit (medical, neuropsychological and experimental) and is lower than 3 months. The study will take place from June 2009 to June 2013.

* Number of patients: 320
* Number of controls: 400
* Potential Benefits expected: criteria for early diagnosis and / or differential diagnosis based on the evaluation process of empathy; elaboration of new clinical tools assisting diagnosis.

ELIGIBILITY:
Inclusion Criteria (Controls):

* being over 18 years old
* speaking French
* in good general health
* affiliated to a welfare state
* given their informed consent in writing

Inclusion Criteria (Patients):

* 18 to 85 years old
* French speaker
* affiliated to a Welfare state
* written consent
* MMSE> 20
* no alexia, agraphia or illiteracy
* absence of diseases that can interfere with cognition (neoplasia, chronic alcoholism ...) of current or past neurological diseases other than those which justified the support nervous system (meningitis, encephalitis, brain injury, developmental disorders, deficits sensory or motor, epilepsy requiring treatment today ...), or of psychiatric disorder (except depression treated)

Exclusion Criteria (controls):

* pathological MMSE score
* insufficient acquisition of the alphabet
* reading, writing, arithmetic
* the presence of a visual deficit or hearing deficit disturbing the tests, paralysis of the dominant hand
* the presence of brain pathology interfering, neurological or psychiatric history

Exclusion Criteria (Patients):

* difficulties in reading, writing or illiteracy
* diseases that can interfere with cognition (neoplasia, chronic alcoholism ...)
* current or past neurological diseases other than those which justified the neurological consultation, Psychiatric pathology (except depression treated)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Empathy ability | 3 months
  Empathy ability is a composite index associating performance on 3 tests (Facial emotion recognition, Theory of Mind and 'Faux pas')

SECONDARY OUTCOMES:
Empathy for pain | 3 months
  pain rating on pictures when others are involved
pattern of empathy disorders according to the disease (stroke, Mild cognitive impairment, Alzheimer disease and Parkinson disease | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Godefroy, PhD-MD, Study Chair — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, Picardie, France

REFERENCES:
- [Result] Narme P, Mouras H, Roussel M, Devendeville A, Godefroy O. Assessment of socioemotional processes facilitates the distinction between frontotemporal lobar degeneration and Alzheimer's disease. J Clin Exp Neuropsychol. 2013;35(7):728-44. doi: 10.1080/13803395.2013.823911. Epub 2013 Aug 12. PMID 23930667
- [Result] Narme P, Mouras H, Roussel M, Duru C, Krystkowiak P, Godefroy O. Emotional and cognitive social processes are impaired in Parkinson's disease and are related to behavioral disorders. Neuropsychology. 2013 Mar;27(2):182-92. doi: 10.1037/a0031522. PMID 23527646